CLINICAL TRIAL: NCT04879966
Title: A Multicenter Prospective Cohort Study Comparing Infliximab to Corticosteroids for Moderate to Severe Ulcerative Colitis
Brief Title: A Cohort Study Comparing IFX to CS for Moderate to Severe UC
Acronym: INSURE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Sponsor
Other Study IDs: 2021ZSLYEC-102
Record Dates: First submitted 2021-05-06; First posted 2021-05-10 (Actual); Last update posted 2022-11-25 (Actual); Status verified 2022-11

CONDITIONS: Moderate to Severe Ulcerative Colitis
MeSH Terms: interventions — Infliximab; Adrenal Cortex Hormones

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- UC cohort: the patiente of Moderate to Severe Ulcerative Colitis who recieved infliximab(IFX) or corticosteroids(CS) as induction therapy would be enrolled in this cohort
  Interventions: Drug: Infliximab; Drug: Corticosteroid

INTERVENTIONS:
Drug: Infliximab — Infliximab was used as induction therapy in UC patients, the maintenance treatment was decided by the researcher
  Other Names: IFX
Drug: Corticosteroid — Corticosteroids was used as induction therapy in UC patients, the maintenance treatment was decided by the researcher
  Other Names: CS

SUMMARY:
The first-line treatment strategy of moderate to severe UC was a important question at issue. The biological agents had potentiality to alter the disease course of UC. The AGA clinical guidelines had conditional recommend that IFX and other biological agene migtht be first-line therapy for high-risk UC patints but only had low grade evidence.We launched this multicenter prospective cohort trial to compare the efficacy and safety of infliximab (IFX) and corticosteroids(CS) when they was used as first-line therapy in UC patients.

ELIGIBILITY:
Inclusion Criteria:

* moderately to severely active ulcerative colitis, defined as a total score of 6 to 12 on the Mayo scale (scores range from 0 to 12, with higher scores indicating more severe disease) and a subscore of at least 2 on the endoscopic component of the Mayo scale (subscores on each of the four components of the Mayo scale range from 0 to 3)
* Patients who had colonic involvement of at least 15 cm
* Patients who had a confirmed diagnosis of ulcerative colitis at least 3 months before screening and confirmed by Pathology

Exclusion Criteria:

* Patients who had previously used any TNF inhibitor
* Patients who were steroid-dependent or steriod-resistant
* Patients who had undergone subtotal colectomy or total colectomy
* Patients who had stoma

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults patinets of moderately to severely active ulcerative colitis who will initiate IFX or CS
Sampling Method: Probability Sample
Enrollment: 342 (Estimated)
Dates: Start 2021-05-17 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
clinical remission | week 14
  defined as a total score of ≤2 on the Mayo scale and no subscore >1; partial Mayo score ≤ 2, no individual subscore > 1

SECONDARY OUTCOMES:
clinical response in induction phase | week 14
  defined as a reduction in the partial Mayo score [stool frequency, rectal bleeding, and physician's global assessment] of ≥2 points and of ≥25% from baseline, with an accompanying decrease in rectal bleeding subscore of ≥1 point or absolute rectal bleeding subscore of ≤1 point
mucosal healing in induction phase | week 14
  defined as a subscore of 0 or 1 on the Mayo endoscopic component
histological healing in induction phase | week 14
  defined as Nancy index score of 0
clinical response in maintenance phase | week 52
  defined as a reduction in the partial Mayo score [stool frequency, rectal bleeding, and physician's global assessment] of ≥2 points and of ≥25% from baseline, with an accompanying decrease in rectal bleeding subscore of ≥1 point or absolute rectal bleeding subscore of ≤1 point
mucosal healing in maintenance phase | week 52
  defined as a subscore of 0 or 1 on the Mayo endoscopic component
histological healing in maintenance phase | week 52
  defined as Nancy index score of 0
quality of life in induction phase | week 14
  defined as an increase of ≥16 points in IBDQ score
quality of life in maintenance phase | week 52
  defined as an increase of ≥16 points in IBDQ score
adverse events | week 52
  as assessed by the incidence of adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- The Sixth Affiliated Hospital, Sun Yat-sen University, Guandong, China